CLINICAL TRIAL: NCT06531447
Title: First-line Gemcitabine Plus Cisplatin in Locally Advanced (IIIC Stage) Breast Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The National Center of Oncology, Azerbaijan (Other Government)
Responsible Party: Principal Investigator, Elchin Mansurov, Head of the Chemothrapy II, The National Center of Oncology, Azerbaijan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOM-0004
Record Dates: First submitted 2024-04-08; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; TUBB3 gene; ERCC1 gene; RMM1 gene; Prognosis and predictive
MeSH Terms: conditions — Breast Neoplasms; Fibrosis Of Extraocular Muscles, Congenital, 3A, with or without Extraocular Involvement | interventions — Cisplatin; Gemcitabine; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Doxorubicin 60mg/m2(Adriblastin) plus Cyclophosphamide 600mg/m2 (endoxan) IV, on 1st days every 3 weeks of 4 cycles. Paclitaxel (Taxol) 80mg/m2, IV every week of 12 cycles or 175mg/m2, IV, on 1st days every 3 weeks of 4 cycles.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel
- Experimental group (Active Comparator): 1250 mg/m2 Gemcitabine 1st and 8th days of 6 cycles and 75mg/m2 Cisplatine 1st day every 3 weeks of 6 cycles
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Cisplatin — Every 21 days 6 cycles
  Other Names: CDDP
  Arms: Experimental group
Drug: Gemcitabine — Every 21 days (First and 8th days) 6 cycles
  Other Names: Gemcitabine hydrochlorid
  Arms: Experimental group
Drug: Doxorubicin — Every 21 days 4 cycles
  Arms: Control group
Drug: Cyclophosphamide — Every 21 days 4 cycles
  Arms: Control group
Drug: Paclitaxel — Every 21 days 4 cycles or once a week for 12 weeks
  Arms: Control group

SUMMARY:
The goal of the study is to investigate of the prognostics and predictive role of TUBB3 expression in locally advanced breast cancer

DETAILED DESCRIPTION:
Using combination of gemcitabine plus cisplatine as first line treatment patients with locally advanced breast cancer with high TUBB3 expression

ELIGIBILITY:
Inclusion Criteria:

IIIC stage breast cancer patients

Exclusion Criteria:

Other stages breast cancer patients

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05; Primary Completion 2017-11 (Actual); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Clinical tumor regression rate | 4 months
  Chemotherapy combination Gemcitabine with Cisplatin

SECONDARY OUTCOMES:
Increasing PFS and OS | 5 years and 10 years
  Observation after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Elchin Mansurov, PhD, Principal Investigator — The National Center of Oncology
Locations (1):
- Elchin Mansurov, Baku, Azerbaijan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Available from 2022
Access Criteria: Breast cancer specialists